CLINICAL TRIAL: NCT04044924
Title: Geriatric Head Trauma Short Term Outcomes Project
Acronym: GREAT-STOP
Status: Completed | Type: Observational
Sponsor: Florida Atlantic University (Other)
Responsible Party: Sponsor
Other Study IDs: 1326154
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-08

CONDITIONS: Head Injury; Anticoagulant-induced Bleeding; Fall
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study will examine the incidence of intracranial hemorrhage. The investigators will compare patients on anticoagulant and/or antiplatelet therapy with head trauma compared to patients not on these medications. While many studies have sought to quantify the incidence of intracranial hemorrhage in these patients, there is considerable controversy regarding their care and what to do after an initial negative head CT in anticoagulated geriatric patients who have experienced head trauma.

ELIGIBILITY:
Inclusion Criteria: Patients seen in the emergency department for head trauma

Exclusion Criteria: Penetrating head trauma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Delray Medical Center and St. Mary's Medical Center emergency departments will be the major focal points for the study. These medical centers are located in Palm Beach County, Florida. Florida has the highest percentage of geriatric patients in the United States and, in particular, Palm Beach County has over 250,000 residents over the age of 65.
Sampling Method: Non-Probability Sample
Enrollment: 5387 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with 14 Day ED Returns | 14 days
  Return visit to ED within 2 weeks
Number of Participants with Primary Intracranial Hemorrhage | initial hospital visit
  ICH on initial head CT scan
Number of Participants with Delayed Intracranial Hemorrhage | 14 days
  ICH on repeat CT scan
Number of Participants with Hospitalizations at 14 days | 14 days
  If patient is admitted for any reason after initial ED visit
Mortality of Participants | 60 days
  Death of patient from any cause at primary visit or up to 60 days from follow-up

SECONDARY OUTCOMES:
New Symptoms | 60 days
  Any new symptoms
Life alterations | 60 days
  Descriptive information from telephone interviews about how patients changed activities after head trauma
New interventions since fall | 60 days
  Additional therapies or intervention instituted after minor head trauma

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shih, MD, Principal Investigator — Florida Atlantic University
Locations (2):
- United States (2):
  - Delray Medical Center, Delray Beach, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: No